CLINICAL TRIAL: NCT03687853
Title: Application of Intrahepatic Arterial Infusion Chemotherapy for Patients With High Risk of Liver Metastases After Pancreatic Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAI PDCA 1.0
Record Dates: First submitted 2018-08-20; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Who Have High CTCs Count in Portal Venous Blood; Liver Metastases
Keywords: Pancreatic ductal adenocarcinoma; arterial infusion chemotherapy; liver metastases

STUDY DESIGN:
Intervention Model Description: Pancreatic cancer patients who received hepatic arterial perfusion chemotherapy after operation
Who Masked: Participant
Masking Description: Pancreatic cancer patients who received chemotherapy through peripheral vein after operation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrahepatic Arterial Infusion chemotherapy (Experimental): chemotherapy through intrahepatic arterial Infusion is one of the most widely used liver tumor treatments.
  Interventions: Device: Intrahepatic Arterial Infusion
- control (No Intervention): chemotherapy through Peripheral venous is one of the regularly used method.

INTERVENTIONS:
Device: Intrahepatic Arterial Infusion — Intrahepatic Arterial Infusion chemotherapy is one of the most widely used liver tumor treatments.
  Arms: Intrahepatic Arterial Infusion chemotherapy

SUMMARY:
Clinical results on intra-arterial adjuvant chemotherapy for prevention

of liver metastasis following curative resection of pancreatic cancer

DETAILED DESCRIPTION:
In this study, the investigator try to select 80 patients who received radical surgery for pancreatic cancer, whose circulating tumor cells(CTCs) count then performed on intraoperative portal venous blood to predict postoperative liver metastasis and were divided into two groups. for those who have high CTCs count may have more chance for the occurrence of postoperative liver metastasis was applied hepatic arterial perfusion chemotherapy with minimal dynamic randomization. The aim is to evaluate the feasibility of hepatic arterial infusion chemotherapy for the prevention of postoperative liver metastasis and improvement of prognosis of pancreatic cancer, so as to further improve postoperative management of pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* pancreatic cancer patients who received the radical operation

Exclusion Criteria:

* who accepted chemotherapy before operation or who cannot or do not will to accepted enrolled into this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | up to 12 months
  Overall survival time after operation

CONTACTS AND LOCATIONS:
Overall Officials: dianrong xiu, doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Department of General Surgery,Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No